CLINICAL TRIAL: NCT00904007
Title: Interactive Spaced Education to Optimize Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EDU 08-422
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: Educational Technology; Hypertension; Education, Professional
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SE Game Cohort (Experimental): Will receive ISE intervention.
  Interventions: Other: Interactive Spaced Education (ISE) --- online education
- Control Cohort (No Intervention): The control cohort will receive identical content online (with no ISE)

INTERVENTIONS:
Other: Interactive Spaced Education (ISE) --- online education — ISE is a novel educational methodology based on the "spacing effect", the psychological finding that repeated presentations of educational material over spaced intervals increase learning efficiency and improve knowledge retention. ISE is delivered using periodic emails that contain clinical case scenarios and multiple-choice questions.
  Arms: SE Game Cohort

SUMMARY:
Online interactive spaced education (ISE) is a novel educational methodology based on the "spacing effect", the psychological finding that repeated presentations of educational material over spaced intervals increase learning efficiency and improve knowledge retention. ISE is delivered using periodic emails that contain clinical case scenarios and multiple-choice question. The investigators recently completed a randomized trial involving 95 VISN 1 primary care providers (PCPs) which demonstrated that an ISE intervention can significantly improve clinician's practice patterns. Those clinicians randomized to the ISE intervention on prostate cancer screening demonstrated a 26% relative reduction in inappropriate screening. The investigators propose to conduct a randomized controlled trial involving PCPs in VISN 1 to determine whether ISE can (1) increase knowledge of the appropriate treatment of hypertensive patients, (2) reduce clinical inertia in hypertension management, and (3) improve the blood pressure control in hypertensive patients.

Anticipated Impacts on Veterans' Healthcare: This study aims to demonstrate that online interactive spaced education (ISE) can improve providers' care of patients with hypertension. ISE is the type of intervention that can be deployed across the VHA with content tailored to meet specific needs and can be implemented as a tool to improve performance measures and clinical outcomes

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans' Healthcare: This study aims to demonstrate that online interactive spaced education (ISE) can improve providers' care of patients with hypertension. ISE is the type of intervention that can be deployed across the VHA with content tailored to meet specific needs and can be implemented as a tool to improve performance measures and clinical outcomes.

Project Background/Rationale: ISE is a novel educational methodology based on the "spacing effect", the psychological finding that repeated presentations of educational material over spaced intervals increase learning efficiency and improve knowledge retention. ISE is delivered using periodic emails that contain clinical case scenarios and multiple-choice questions. We recently completed a randomized trial involving 95 VISN 1 primary care providers (PCPs) which demonstrated that an ISE intervention can significantly improve clinician's practice patterns. Those clinicians randomized to the ISE intervention on prostate cancer screening demonstrated a 26% relative reduction in inappropriate screening.

Project Objectives: Lowering blood pressure in hypertensive patients unequivocally decreases the incidence of stroke and cardiovascular events and is highly cost-effective. The majority of patients with blood pressure above the treatment target do not have their anti-hypertensive medications appropriately intensified at clinician visits. A reduced frequency of treatment intensification is alternatively termed 'clinical inertia'. Our preliminary results show that clinicians' knowledge of hypertension management guidelines is limited, and few clinicians report following the guidelines consistently. We propose to conduct a randomized controlled trial involving PCPs in VISN 1 to determine whether ISE can (1) increase knowledge of the appropriate treatment of hypertensive patients, (2) reduce clinical inertia in hypertension management, and (3) improve the blood pressure control in hypertensive patients.

Project Methods: One hundred six VISN 1 primary care practitioners (physicians, nurse practitioners, and physician assistants) will be recruited via email to participate in the study. Participants will be randomized to one of two cohorts: (1) the intervention cohort will receive ISE over year 1, and (2) the control cohort will receive no intervention and will represent the "standard of education" on hypertension management. The ISE intervention will consist of an email every 4 days containing 1 multiple-choice questions based on a curriculum derived from clinical practice guidelines on appropriate hypertension management. Providers will submit answers to the questions online and immediately receive the correct answer and an explanation of the pertinent clinical issues. Using a new adaptive methodology, the spacing and content of the educational intervention will be individualized for each clinician based on their performance. The ISE intervention will be completed in 9-11 months. Hypertension knowledge will be assessed by a post-test at the end of year 1. Providers' clinical inertia and the blood pressures of their patients will be assessed over 2 years: initial changes attributable to ISE will be identified in year 1, while the retention of these changes will be monitored in year 2. Drawing on the interdisciplinary expertise of our investigator team, the study is positioned to enrich national debates about how best to improve the ways in which clinicians can meet their lifelong learning needs.

ELIGIBILITY:
Inclusion Criteria:

* VA VISN 1 primary care clinicians (MD, NP, PA) who have at least a 50% (4/8 time) clinical appointment.

Exclusion Criteria:

* VA VISN 1 primary care clinicians (MD, NP, PA) who do not have at least a 50% (4/8 time) clinical appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Price Kerfoot, MD EdM, Principal Investigator — VA Boston Healthcare System Brockton Campus, Brockton, MA
Locations (1):
- VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts, United States

REFERENCES:
- [Result] Kerfoot BP, Turchin A, Breydo E, Gagnon D, Conlin PR. An online spaced-education game among clinicians improves their patients' time to blood pressure control: a randomized controlled trial. Circ Cardiovasc Qual Outcomes. 2014 May;7(3):468-74. doi: 10.1161/CIRCOUTCOMES.113.000814. PMID 24847084

RESULTS

PARTICIPANT FLOW:
Groups:
- SE Game Cohort: SE game clinicians were e-mailed one question every 3 days. Adaptive game mechanics re-sent questions in 12 or 24 days if answered incorrectly or correctly, respectively. Clinicians retired questions by answering each correctly twice consecutively. Posting of relative performance among peers fostered competition.
- Control Cohort: Control clinicians received identical educational content in an online posting with email reminders.
Period: Overall Study
Arm/Group | SE Game Cohort | Control Cohort
Started | 55 | 56
Completed | 55 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants' baseline demographic characteristics were similar between randomized cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | SE Game Cohort | Control Cohort | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (9.7) | 53.1 (8.5) | 51.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cross-cohort Comparison of the Average Time Needed to Normalize Patients' Blood Pressure
Description: A unique hypertensive period served as the unit of analysis. A hypertensive period started on the first day during the study when a patient's BP was elevated. It ended on the first subsequent day when it was <140/90 mm Hg or on the last day BP was recorded during the study. Duration of the hypertensive period (days) was the outcome measure. BP measurements obtained in the course of routine care were used to ascertain study outcomes, whether obtained by the PCP or at other clinic visits. These measurements were obtained from structured data (ie, BP recordings in the electronic medical record) and natural language processing of provider notes as previously described. If several measurements were recorded on the same day, the lowest mean arterial BP was used.
Time Frame: Months 1-24
Measure: Median (Full Range); unit: days
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 55 | 56
days | 137 [0 to 365] | 145 [0 to 365]

2. Secondary Outcome: Cross-cohort Comparison of Patients' Average Blood Pressure at 12 Months After Trial Launch (Last Measured Blood Pressure in Months 1-12)
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cross-cohort Comparison of Patients' Average Change in Blood Pressure Over Months 1-12 (Last Measured Blood Pressure in Months 1-12)
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cross-cohort Comparison of Patients' Average Blood Pressure at 24 Months After Trial Launch (Last Measured Blood Pressure in Months 13-24)
Time Frame: Months 13-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cross-cohort Comparison of Patients' Average Change in Blood Pressure Over Months 13-24 (Last Measured Blood Pressure in Months 13-24)
Time Frame: Months 13-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cross-cohort Comparison of Patients' Average Blood Pressure at 24 Months After Trial Launch (Last Measured Blood Pressure in Months 1-24)
Time Frame: Months 1-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Cross-cohort Comparison of Patients' Average Change in Blood Pressure Over Months 1-24 (Last Measured Blood Pressure in Months 1-24)
Time Frame: Months 1-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cross-cohort Comparison of Frequency of Treatment Intensification
Time Frame: Months 1-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Cross-cohort Comparison of Patients' Follow-up Intervals After Clinical Encounters With Elevated Blood Pressure
Time Frame: Months 1-24
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Pre-test Performance Differences by Provider-related Variables (Site of Care, Age, Date of Recertification, Etc.)
Time Frame: Month 1
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Cross-cohort Comparison of Providers' Post-test Scores (Score Improvements)
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Baseline Knowledge Levels of Providers Assessed Via Their Initial Responses to Spaced Education Items (Spaced Education Cohort Only)
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Performance Differences by Provider-related Variables (Site of Care, Age, Date of Recertification, Sex, Etc.) in the Spaced Education Program (Spaced Education Cohort Only)
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Provider-perceived Acceptability of Spaced Education Intervention
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Provider-perceived Effectiveness of Spaced Education Intervention
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Providers' Perceptions of the Optimal Parameters for the Spaced Education Intervention
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Provider-perceived Barriers and Facilitators to the Spaced Education Intervention
Time Frame: Months 1-12
Population: PI and project staff no longer have access to the raw data and are no longer able to generate any more data analyses.
Arm/Group | SE Game Cohort | Control Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm 1: SE game clinicians were e-mailed one question every 3 days. Adaptive game mechanics re-sent questions in 12 or 24 days if answered incorrectly or correctly, respectively. Clinicians retired questions by answering each correctly twice consecutively. Posting of relative performance among peers fostered competition.
- Arm 2: Control clinicians received identical educational content in an online posting with email reminders.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No